CLINICAL TRIAL: NCT04469413
Title: Comparison of The Effect of Continuous and Standard Intermittent Boluses Paracetamol Infusion on Patent Ductus Arteriosus
Brief Title: Comparison of Infusion Paracetamol Protocols in PDA
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ufuk Cakir, Ankara University, Ankara University
Other Study IDs: 113/2019
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Patent Ductus Arteriosus in Preterm Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard IV intermittent bolus infusion group
  Interventions: Drug: Paracetamol Infusion
- continuousIV intermittent bolus infusion group
  Interventions: Drug: Paracetamol Infusion

INTERVENTIONS:
Drug: Paracetamol Infusion — Continuous and Standard Intermittent Boluses Paracetamol Infusion

SUMMARY:
The aim of this study was to evaluate the effect of paracetamol on patent ductus arteriosus (PDA) closure and clinical outcomes in preterm infants when used as standard intermittent bolus and continuous intravenous (IV) infusion. Preterm neonates with birth weight (BW) ≤1500 g and gestational age (GA) ≤32 weeks were included in this study. During the study period, IV paracetamol therapy was given to all infants with hemodynamically significant patent ductus arteriosus (hsPDA). The patients were divided into the standard IV intermittent bolus infusion group and the continuous IV infusion group.

DETAILED DESCRIPTION:
Demographic and clinical features Perinatal variables were recorded for all infants, including GA, BW, sex, APGAR scores (at 1 and 5 minutes), prenatal steroids, pre- and post-treatment alanine aminotransferase (ALT)/aspartate aminotransferase (AST), second and third courses of paracetamol, PDA ligation, clinical variables including respiratory distress syndrome (RDS), IVH (grade ≥3), NEC (grade≥2), moderate or severe BPD, ROP requiring laser therapy, early-onset neonatal sepsis (EOS), late-onset sepsis (LOS), duration of non-invasive ventilation (NIV), mechanical ventilation (MV) and oxygen (O2) supplementation, day of full enteral feeding achievement, length of hospital stay, and mortality.

Sepsis with onset at ≤72 hours was defined as EOS and at >72 hours as LOS in infants hospitalized in the NICU. RDS was defined as the need for surfactant administration [5]. IVH was diagnosed by cranial ultrasound in the first 7 days of life (intraparenchymal hemorrhage + IVH, large IVH). NEC diagnosis and staging were implemented by using Bell's criteria. Neonates that received positive pressure or ≥30% oxygen without pressure after a postmenstrual age of 36 weeks were diagnosed as having moderate or severe BPD [8]. ROP screening was done by ophthalmologists according to the International Classification of Retinopathy of Prematurity Revisited [9].

Hemodynamically Significant Patent Ductus Arteriosus All neonates underwent Doppler echocardiography (ECHO) at postnatal 72 hours. Diagnosis of hsPDA was based on clinical and ECHO features [10]. ECHO evaluation was repeated at regular intervals. IV paracetamol was used as primary rescue therapy for hsDPA. If hsPDA persisted despite 3 courses of paracetamol therapy, surgical ligation was performed. The non-hsPDA group comprised non-hsPDA preterm infants selected using the same exclusion criteria. Infants with non-hsPDA were excluded from the study.

Continuous and Standard Intermittent Bolus Infusion of Paracetamol IV paracetamol therapy was delivered as primary rescue pharmacological treatment to all neonates who had hsPDA during the study period. Standard IV intermittent bolus paracetamol therapy was administered in the form of 15 mg/kg doses as 1-hour infusions every 6 hours for 5 days, while continuous IV paracetamol infusion therapy was administered as a 60 mg/kg/day dose continuously for 5 days (Parol, Atabay Ilac Kimya San., Istanbul, Turkey). ALT and AST levels were analyzed before and after treatment . Infants received standard IV intermittent bolus paracetamol between January 1 and April 31, 2018, and continuous IV infusion paracetamol between May 1 - August 31, 2018 for hsPDA medical treatment. Therefore, eligible infants were divided into two groups as the standard IV intermittent bolus infusion group and the continuous IV infusion group.

ELIGIBILITY:
Inclusion Criteria:

birth weight (BW) ≤1500 g and gestational age (GA) ≤32 weeks at birth

Exclusion Criteria:

birth weight (BW) >1500 g and gestational age (GA) >32 weeks at birth

Max Age: 1 Month | Sex: All
Age Groups: Child
Study Population: Preterm preterms with birth weight (BW) ≤1500 g and gestational age (GA) ≤32 weeks will be included in the study.
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Patent Ductus Arteriosus | 6 months
  PDA-related morbidities, multiple paracetamol courses, and PDA ligation

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk Cakir, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cakir U, Tayman C, Karacaglar NB, Beser E, Ceran B, Unsal H. Comparison of the effect of continuous and standard intermittent bolus paracetamol infusion on patent ductus arteriosus. Eur J Pediatr. 2021 Feb;180(2):433-440. doi: 10.1007/s00431-020-03822-1. Epub 2020 Sep 29. PMID 32995919